CLINICAL TRIAL: NCT03551470
Title: Robot-assisted Resection of Colorectal Cancer and Synchronous Liver Metastases:Preliminary Experience, Technique and Literature Review
Brief Title: Minimally Invasive Simultaneous Colorectal and Liver Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera San Giovanni Battista (Other)
Responsible Party: Principal Investigator, Michele De Rosa, Principal Investigator, Azienda Ospedaliera San Giovanni Battista
Other Study IDs: AOSGB1
Record Dates: First submitted 2018-05-28; First posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Colorectal Cancer
Keywords: robotic; laparoscopy; liver surgery; colorectal and synchronous liver metastases; simultaneous surgery
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Synchronous colorectal cancer and liver metastases: Robotic (Da Vinci) one-stage colorectal and liver resection
  Interventions: Procedure: Robotic one-stage colorectal and liver resection

INTERVENTIONS:
Procedure: Robotic one-stage colorectal and liver resection

SUMMARY:
Up to 25% of newly diagnosed patients with colorectal cancer (CRC) have liver metastases (LM). Simultaneous colorectal and hepatic resection has been proven to be a safe and effective approach in dealing with metastatic colorectal cancer.

The aim of this paper is to analyse perioperative and oncological outcomes of minimally invasive (laparoscopic and robotic) one-stage simultaneous resection of liver metastases and colorectal tumor in selected patients affected by colorectal cancer and synchronous liver metastases.

DETAILED DESCRIPTION:
From October 2012 to March 2018 a minimally invasive one-stage resection was offered to selected patients referred to the investigator's institution with a diagnosis of CRC and synchronous LM, irrespective of the size and location of the primary and metastatic disease. When feasible, a fully-robotic colorectal and liver resection was performed. Prior consent was obtained and full treatment options where submitted to all patients treated. Data collected were prospectively analyzed.

Diagnosis and pre-operative staging were achieved with pancolonoscopy with biopsies and, where contraindicated or not feasible, with CT colonography.

Pelvic MRI with rectal cancer protocol was used for local staging of rectal cancer and total-body contrast-enhanced computed tomography (CT) and liver contrast-enhanced magnetic resonance imaging (MRI) for investigation of metastases. In selected cases a CEUS (contrast-enhanced ultrasound) or liver biopsy was performed in order to achieve a diagnostic definition.

All cases were discussed at multidisciplinary team meeting. Criteria for neoadjuvant chemotherapy were liver unresectability with a potential incomplete liver resection with anticipated positive surgical margins and an insufficient liver remnant.

Absolute contraindications for minimally invasive simultaneous surgery were considered unfitness for surgery due to comorbidities not allowing long operative time, the number of lesions in parenchymal sparing surgery (generally >5), the pre-operative prediction of vascular resection.

Relative contraindications were considered the need for major hepatectomy and the finding of new intraoperative lesions, with consequent potential longer operative time.

Demographic, histopathological, surgical morbidity/mortality and short term peri-operative clinical outcome in all patients undergone simultaneous colorectal and liver resections were prospectively evaluated.

Morbidity evaluation included all intra-operative and early post-operative (within 30 days) complications and rated according to Clavien-Dindo classification.

All data are expressed as mean values ± range when appropriate

ELIGIBILITY:
Inclusion Criteria:

* colorectal primary tumor with synchronous liver metastases
* eligibility for minimally-invasive surgery

Exclusion Criteria:

* unfitness for prolonged operative time
* liver lesions >5
* pre-operative prediction of vascular resection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Selected patients affected by colorectal cancer with synchronous liver metastases
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2012-10 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Short-term perioperative surgical outcomes | intra-operative - within 30 post-operative day
  Morbidity
Mortality | Intra-operative -within 30 post-operative day
Blood loss | Intra-operative
  Measured in mL
Conversion rate | Intra-operative
Operative time | Intra-operative
  Measured in minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Michele De Rosa, Foligno, Perugia, Italy

IPD SHARING:
Plan to Share IPD: Undecided